CLINICAL TRIAL: NCT03744325
Title: Humoral and Cellular Immune Responses in Hen's Egg Oral Immunotherapy
Brief Title: Immune Responses in Hen's Egg Oral Immunotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Kati Palosuo, MD, PhD, Principal investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HOIT01
Record Dates: First submitted 2018-11-12; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Food Allergy; Egg Protein Allergy; Immune Tolerance
Keywords: Food allergy; Hen's egg allergy; Desensitization; Oral immunotherapy (OIT); Systems biology
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Patients are randomized 2:1 to receive active HE OIT or continue on an elimination diet after which active HE OIT is started.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hen's egg OIT (Active Comparator): Daily intake of gradually increasing doses of egg white protein under a 32 weeks period, continued by regular, daily intake of 1000 mg egg white protein.
  Interventions: Dietary Supplement: Hen's egg OIT
- Hen's egg avoidance (No Intervention): Hen's egg is avoidance diet is continued.

INTERVENTIONS:
Dietary Supplement: Hen's egg OIT — Increasing doses of egg white protein administered orally
  Arms: Hen's egg OIT

SUMMARY:
The study determines how a 6 months oral immunotherapy (OIT) program with hen's egg (HE) effects cellular and humoral immune responses in 50 children with HE allergy. Clinical data, transcriptomics and epigenetics are combined and analyzed by advanced system biology methods. This study will provide better understanding of the effects and mechanisms of OIT.

DETAILED DESCRIPTION:
Oral immunotherapy (OIT) is a therapeutic approach, where gradually increasing doses of a specific food allergen are administered orally. OIT can desensitize up to 80% of children with persistent food allergy, and in a subset lead to sustained immune tolerance. The immunologic mechanisms induced by OIT are still poorly understood.

In this randomized cross-over study, 50 children with challenge-confirmed hen's egg (HE) allergy will be randomized (2:1) to receive either active HE OIT or continue on an avoidance diet for 6 months after which active OIT is started. The immunological changes induced by OIT will be compared to the patient's initial status and to that of the patients on an avoidance diet.

Serum antibody and humoral mediator analyses as well as gene expression of blood mononuclear cell (PBMC) by genome-wide microarray assays will be studied. PBMCs will be stimulated with HE allergens and innate immunity agonists, and the differences in the expression profiles of messenger-RNAs as well as microRNAs will be studied. Single-cell sequencing and sorting of regulator T cells (Tregs) will be performed focusing on their transcriptomic responses and gene methylation. Finally, clinical data, transcriptomics and epigenetic changes will be combined and analyzed by advanced system biology methods.

This study will provide better understanding of the effects and mechanisms of OIT and identify biomarkers for selection of patients benefitting from personalized OIT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-19 years
2. Sensitization to egg white (egg white- specific IgE ≥0.35 kU/l or skin prick test ≥3 mm)
3. Positive double-blind, placebo-controlled food challenge to heated egg white

Exclusion Criteria:

1. Poor adherence
2. Uncontrolled or severe asthma
3. Severe systemic illness
4. Active autoimmune disease
5. Active, malignant neoplasia

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03-18 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
OIT-induced allergen-specific antibody responses | Up to 32 weeks
  The amount of specific serum IgE, IgG4, and IgA antibodies (kU/L) to the major egg allergens (Gal d1 - d4) will be measured by ImmunoCAP after 0, 14, and 32 weeks of OIT or avoidance.
OIT-induced changes in the peripheral blood cell transcriptome | Up to 32 weeks
  Gene expression of blood mononuclear cells (PBMC) after 0, 14 and 32 weeks of OIT or avoidance will be studied. Total-RNA extracted from PBMCs will be used for microarrays. The genome-wide expression of the approximately 25.000 genes will be investigated on Agilent SurePrint G3 Human Gene Expression v3 arrays.
OIT-induced allergen-specific expression profiles of messenger-RNAs and microRNAs | Up to 32 weeks
  Comprehensive highthroughput sequencing for long (mRNA) and short (miRNA) coding gene expression approach will be used to investigate transcriptional changes in exposed blood cells after different stimulations (egg extract, LPS, PolyI:C)

SECONDARY OUTCOMES:
The prorportion of participants able to consume 1000mg of egg protein after 32 weeks of OIT | Up to 32 weeks
  Measured in mg of egg protein consumed without symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Mika J Mäkelä, Professor, Study Director — Skin and Allergy Hospital, Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: Undecided